CLINICAL TRIAL: NCT03441672
Title: Improved Prenatal Genetic Screening Decision Making Through Interactive Technology
Brief Title: Game-Based Decision Aid to Educate Pregnant Women About Prenatal Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R21HD083832 (NIH); R21HD083832 (NIH)
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Prenatal Disorder
Keywords: Prenatal Screening; Interactive educational technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group interact with the game technology to learn about prenatal screening, in addition to usual care provided in the clinic.
  Interventions: Behavioral: Meaning of Screening
- Control (No Intervention): Participants in the control group learn about prenatal screening through usual care in the clinic.

INTERVENTIONS:
Behavioral: Meaning of Screening — Interactive technology game providing education about prenatal screening and what the results may mean.
  Arms: Intervention

SUMMARY:
Significant barriers exist for effectively informing women about prenatal screening in the clinical setting. This project developed and evaluated the efficacy of a game decision aid among pregnant women about prenatal screening in a randomized controlled study.

DETAILED DESCRIPTION:
Prenatal genetic screening has grown at a rapid rate and whole genome sequence of an unborn fetus is expected to be widely available in the next few years. However, significant barriers remain for effectively informing couples about their risks and options for identifying and managing chromosomal anomalies and heritable conditions during pregnancy. It is widely recognized that current standards for patient education in this domain are largely ineffective. Decisions about prenatal screening are based on pregnant couples' values and knowledge so clinicians are often challenged with being informative but non-directive. Prenatal screening has grown significantly in recent years because the American College of Obstetricians and Gynecologists recommends prenatal care providers now offer all women prenatal genetic screening in the first trimester of pregnancy, regardless of age, or genetic risk status. This has moved the focus of prenatal screening from a subset of higher risk pregnant couples to all pregnant couples and to an earlier time in pregnancy.

To address these information needs, we are undertaking a novel approach to inform couples about screening. "Gaming" tools have demonstrated promising outcomes for improved health care decision-making and compliance with health recommendations. In contrast to other computer applications for the dissemination of information, game technology goes beyond information delivery and engages users in different life choice scenarios. Further, these tools can assess whether the attractiveness (or unattractiveness) of different simulated choices can offer insights about one's values. In this value-laden context, the game allows individuals to explore their personal values in a non-directive fashion and allows a comparison of the game choices and values with an individual's reproductive partner.

The purpose of this application is to 1) develop a prenatal screening gaming application prototype (PS-GAP) and 2) conduct a preliminary assessment of the PS-GAP on knowledge, satisfaction, and decisional conflict about prenatal genetic screening for pregnant women and their partners.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* less than 15 weeks gestation
* attending first obstetric visit
* low risk pregnancy

Exclusion Criteria:

* Non-English speaking
* High risk pregnancy
* Past 15 weeks gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Level of knowledge about prenatal screening and prenatal diagnostic testing | Immediately after intervention
  prenatal screening knowledge is measured with a 23-item survey developed by an expert panel of genetic counselors, physicians, social scientists and data collection experts. All questions use a five point likert scale for response.

SECONDARY OUTCOMES:
Documentation of decision to undergo prenatal screening | Up to 4 weeks after intervention
  Documentation of participant's decision to complete prenatal screening or not, as pulled from the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rothwell, PhD, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared, only unidentified aggregate data.